CLINICAL TRIAL: NCT04233268
Title: RASCALS: Rapid Assay for Sick Children With Acute Lung Infection Study
Acronym: RASCALS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Cambridge University Hospitals NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Dr Nazima Pathan, University Lecturer in Paediatric Intensive Care, Cambridge University Hospitals NHS Foundation Trust
Other Study IDs: 277039
Record Dates: First submitted 2020-01-15; First posted 2020-01-18 (Actual); Last update posted 2021-10-20 (Actual); Status verified 2021-10

CONDITIONS: Lower Respiratory Tract Infection; Ventilator Associated Pneumonia; COVID19
MeSH Terms: conditions — Pneumonia, Ventilator-Associated; COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Bronchoalveolar Lavage fluid, Blood
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Critically ill children: Children with severe infection requiring mechanical ventilation
  Interventions: Diagnostic Test: Rapid Pathogen Detection
- Non critically ill cohort: Children with severe infection admitted to hospital but not requiring mechanical ventilation
- Profiling of the respiratory microbiome: Mechanically ventilated children of any cause admitted to PICU
  Interventions: Diagnostic Test: Rapid Pathogen Detection

INTERVENTIONS:
Diagnostic Test: Rapid Pathogen Detection — Rapid assays for pathogen detection on bronchoalveolar lavage fluid
  Groups: Critically ill children; Profiling of the respiratory microbiome

SUMMARY:
Lower Respiratory Tract infections are a common cause of admission to the intensive care unit. Children routinely receive antibiotics until the tests confirm whether the infection is bacterial or viral. The exclusion of bacterial infection may take 48 hours or longer for culture tests on biological samples to be completed. In many cases, the results may be inconclusive or negative if the patient has already received antibiotics prior to the sample being taken.

A rapid assay to detect the most likely cause of infection could improve the speed with which antibiotic therapy is rationalised or curtailed.

This study aims to assess whether a new genetic testing kit which can identify the presence of bacteria and viruses within hours rather than days is a feasible tool in improving antibiotic prescribing and rationalisation of therapy in critically ill children with suspected lower respiratory tract infection.

ELIGIBILITY:
Inclusion Criteria:

1. Aged >37 weeks corrected gestation and ≤16 years old
2. Receiving mechanical ventilation
3. Commencing or already receiving antibiotic treatment for lower respiratory tract infection

Exclusion Criteria:

1. Survival not expected/active medical treatment expected to be withdrawn/palliative care only

Ages: 0 Months to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Critically ill children with suspected lower respiratory tract infection
Sampling Method: Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2020-06-06 (Actual); Primary Completion 2023-02-28 (Estimated); Study Completion 2025-02-28 (Estimated)

PRIMARY OUTCOMES:
Performance of the novel pathogen detection assay | 3 years
  Performance of novel pathogen detection assays compared to standard microbiology, in regard to sensitivity, specificity and likelihood ratios

SECONDARY OUTCOMES:
Time to results | 3 years
  Time to reportable test results
Negative cultures | 3 years
  Where routine culture is negative, what proportion of tests have a positive detection using the novel assay?
Antibiotic therapy | 3 years
  Duration of therapy and number of antibiotic classes during paediatric intensive care unit admission

OTHER OUTCOMES:
Prevalence of COVID19 in children admitted to PICU | 2 years
  Number of critically ill children requiring mechanical ventilation with COVID19 compared to those without
Prevalence of SARS-CoV-2 antigen in faecal samples following acute admission with COVID-19 related illness | 2 years
  Faecal excretion of SARS-CoV-2

CONTACTS AND LOCATIONS:
Overall Officials: Nazima Pathan, FRCPCH PhD, Principal Investigator — Cambridge University Hospitals NHS Foundation Trust
Locations (1):
- Addenbrooke's Hospital, Cambridge, Cambs, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Clark JA, Conway Morris A, Kanaris C, Inwald D, Butt W, Osowicki J, Schlapbach LJ, Curran MD, White D, Daubney E, Agrawal S, Navapurkar V, Torok ME, Baker S, Pathan N. A qualitative investigation of paediatric intensive care staff attitudes towards the diagnosis of lower respiratory tract infection in the molecular diagnostics era. Intensive Care Med Paediatr Neonatal. 2023;1(1):10. doi: 10.1007/s44253-023-00008-z. Epub 2023 Jul 7. PMID 37425493
- [Derived] Clark JA, Kean IRL, Curran MD, Khokhar F, White D, Daubney E, Conway Morris A, Navapurkar V, Bartholdson Scott J, Maes M, Bousfield R, Gouliouris T, Agrawal S, Inwald D, Zhang Z, Torok ME, Baker S, Pathan N. Rapid Assay for Sick Children with Acute Lung infection Study (RASCALS): diagnostic cohort study protocol. BMJ Open. 2021 Nov 29;11(11):e056197. doi: 10.1136/bmjopen-2021-056197. PMID 34845080